CLINICAL TRIAL: NCT01534104
Title: Using Functional MRI and Diffusion Imaging of Eloquent Brain Areas to Optimize Brain Tumor Resection Planning
Brief Title: MRI and Diffusion Imaging of Eloquent Brain Areas to Optimize Brain Tumor Resection Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-008
Record Dates: First submitted 2012-02-09; First posted 2012-02-16 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Brain Cancer
Keywords: fMRI; DTI; DSI; tractography; neurological/physical testing; Motor and Language Pathways; resting state fMRI; 12-008
MeSH Terms: conditions — Brain Neoplasms; Neurologic Manifestations

ARMS (1):
- pts who have primary or secondary brain tumors (Experimental): The study will prospectively enroll subjects who have primary or secondary brain tumors located near the motor pathway (corticospinal tract) or language pathway (arcuate fasciculus). This is a nonrandomized study in which each subject will receive the standard of care as per the treating neurosurgeon.
  Interventions: Procedure: preoperative fMRI. DTI and DSI with tractography

INTERVENTIONS:
Procedure: preoperative fMRI. DTI and DSI with tractography — W/I approx 4-6 weeks of the fMRI, DTI & DSI, neurological/physical testing & brain MRI showing tumor &/or edema located in or near (<2 cm) the motor cortex (precentral gyrus), motor pathway (corticospinal tract), language cortex (Broca's area, Wernicke's area), &/or language pathway (arcuate fasciculus) Preoperative MRI for surgical planning (approximately <48 hours before surgery*) fMRI to localize gray matter DTI, DSI & tractography to localize white matter, DSI & updated fMRI (Optional) Most patients will undergo surgery w/i 48 hrs of their preoperative MRI. For some patients, the MRI results will be used for preoperative counseling. In this subset of patients, we expect that surgery will occur w/i 3-4 months of the MRI. Brain tumor resection as per the treating neurosurgeon Electrical stimulation to localize gray &/or white matter structures if clinically necessary according to the standard of care at MSKCC Postoperative neurological/physical examination (<48 hours after surgery)

SUMMARY:
Many patients with brain tumors require surgery. Some patients have brain tumors near important parts of the brain. These brain areas have roles in language or motor function. Avoiding these motor and language areas helps to prevent neurological deficits. The investigators are studying the parts of the brain involved in motor and language. Patients usually get functional MRI (fMRI) or resting-state fMRI (rs-fMRI) for gray matter mapping and diffusion tensor imaging (DTI) or diffusion spectrum imaging (DSI) for white matter mapping. These special MRI sequences are used to plan surgery. Patients are scheduled to have imaging to help plan for possible surgery.

Some patients may require stimulation during surgery to motor and language areas. In patients who require stimulation as part of their standard of care, the investigators will compare the investigators imaging results with the stimulation results. The purpose of this study is to improve MRI mapping of the motor and language pathways in the brain.

The scans are necessary stimulation for this protocol are part of the standard of care. In other words, these tests are done as part of the best possible care even if they did not join this study. The investigators are studying new techniques for analyzing the MRI data. These new techniques may give the doctor a better view of where the brain tumor is located relative to important parts of the brain.

The investigators will only perform the test sequences that are necessary for mapping the tumor. Most patients will require both fMRI and DTI. Some patients may only require fMRI or DTI. The investigators may also ask to perform optional sequences during the scan. Multi-echo is an modified form of fMRI. DSI is a modified form of DTI. These optional sequences are for research only. The patient would not get these sequences if they do not enroll in this study.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary brain tumor (enhancing mass lesion ± nonenhancing abnormality), known or suspected, located near (< 2 cm) any portion of the motor cortex, motor pathway, language cortex, or language pathway as determined on anatomical images;
* Planned resection of the tumor;
* fMRI and/or DTI required for preoperative imaging as part of the standard of care
* Patient and/or guardian is able to provide written informed consent prior to study registration
* Age ≥ 18 years old

Exclusion Criteria:

* Unable to tolerate MRI and/or perform fMRI tasks (e.g., severe claustrophobia or pacemaker or aneurysm clip that precludes MRI scan)
* Pregnant or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
standard vs. probabilistic tractography | 1 year
  The standard and probabilistic tractography results will be compared to expected anatomy as determined by expert operators. The reconstructed tracts will be examined for their configurations near the tumor and/or edema, and the completeness of their courses. All analyses will be scored by two expert operators (2 board certified radiologists who hold Certificates of Added Qualification in Neuroradiology and are familiar with DTI and tractography), with disagreements resolved by consensus.

SECONDARY OUTCOMES:
the utility of diffusion spectrum imaging (DSI) | 2 years
  (Optional) DSI is a newly proposed modification of DTI that allows potentially improved visualization of the complex white matter architecture. Recent technical advances have allowed marked reduction of the DSI scan time to match other clinical scan times. DSI in brain tumor patients has not been described Analysis of the DSI results will be performed in a manner similar to the analysis for DTI in Specific Aim #1. Briefly, the endings of the rostral language tracts will be graded as: 0-none; 1-few; 2-some; or 3-all for tracts extending to the fMRI activated Broca's area. Both motor and language tracts will be compared to the contralateral mirror tract using a similar 0-3 scale (0-absent, 3-normal) by two expert operators with disagreements resolved by consensus.
feasibility of updated fMRI sequences | 2 years
  (Optional) rs-fMRI is a newly proposed technique to map functional networks in the brain with data obtained during a quiet, resting state condition - as opposed to the usual task-based fMRI that requires patient cooperation and performance. This is an exploratory aim and no statistical analyses are expected to be performed. We anticipate that all of the patients who undergo rs-fMRI will be able to lie still for the additional approximate 7 min required to acquire the updated fMRI sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Young, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/